CLINICAL TRIAL: NCT06139276
Title: Outcomes of a Specially Designed Needle (Small Needle-Knife) Treating Frozen Shoulder Based on Analysis of Microcirculation and Pulse Changes
Brief Title: Outcomes of Frozen Shoulder Treated With Small Needle-Knife Through Microcirculation and Pulse Analysis.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Taipei City Hospital (Other Government)
Collaborators: National Taiwan University of Science and Technology (Other); National Yang Ming Chiao Tung University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TCHIRB-11206008
Record Dates: First submitted 2023-11-14; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Frozen Shoulder
Keywords: Frozen Shoulder; Acupotomy; Small Needle-Knife; Adhesive Capsulitis; Laser Doppler Flowmetry; Photoplethysmography; Blood Pressure Waveform
MeSH Terms: conditions — Bursitis | interventions — Acupuncture Therapy

STUDY DESIGN:
Intervention Model Description: This study plans to collect 120 individuals diagnosed with frozen shoulder by both Western and Traditional Chinese medicine practitioners, randomized in a 1:1 ratio to receive either standard treatment or a combination of small needle-knife therapy and standard treatment.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Small Needle-Knife (Experimental): The small needle-knife (SNF) group undergoes rehabilitation treatment, with additional small needle-knife treatment once a week after acupuncture needle insertion at the Tiaokou (ST38) and Chengshan (BL57) acupoints. This treatment regimen will span over a duration of 3 weeks.
  Interventions: Procedure: Small Needle-Knife
- Standard treatment (Active Comparator): Rehabilitation treatment (based on the physician's assessment of the patient's clinical condition, using methods such as heat therapy, electrotherapy, manual therapy, or joint injections) at least once a week. This treatment regimen will span over a duration of 3 weeks.
  Interventions: Other: Standard treatment

INTERVENTIONS:
Procedure: Small Needle-Knife — The small needle-knife therapy originated from the ancient Chinese acupuncture instrument known as the "Pi needle" from the "Nine Needles," which resembled a sword, had two sharp edges, and was originally used for abscess drainage. It is currently widely applied in treating conditions such as myofascial adhesions, chronic pain, or nerve compression.
  The small needle-knife features a flat and rounded tip design, with its handle made of solid steel. This construction provides excellent toughness and flexibility, minimizing tissue damage, and facilitating microadhesiolysis, an intervention aimed at releasing adhesions.
  Other Names: Acupotomy
  Arms: Small Needle-Knife
Other: Standard treatment — Standard treatment
  Arms: Standard treatment

SUMMARY:
The aim is to investigate whether adding small needle-knife therapy to standard Western medicine enhances the treatment of frozen shoulder by evaluating its impact on microcirculation and meridian unblocking.

DETAILED DESCRIPTION:
The aim of this research is to investigate whether the combination of small needle-knife therapy with conventional Western medicine treatment can enhance therapeutic effects compared to conventional treatment methods. In addition to clinical measurements of joint mobility and relevant scales, this study integrates instruments such as Laser Doppler Flowmetry (LDF) and pulse diagnosis devices. These non-invasive methods are employed to evaluate the microcirculation performance of patients with frozen shoulder before and after conventional Western medicine treatment or combined treatment with small needle-knife therapy. The objective is to understand the effects of small needle-knife therapy on the microcirculation and meridian unblocking in frozen shoulder patients.

ELIGIBILITY:
Inclusion Criteria:

* Limited shoulder joint mobility in various angles (forward flexion, abduction, external rotation, and internal rotation), persisting for over two months.
* Persistent pain on the affected shoulder even without rest.
* Willing and consenting to participate in this research.

Exclusion Criteria:

* Degenerative shoulder joint arthritis (osteoarthritis).
* Rheumatoid arthritis.
* Fracture of the humerus, clavicle, scapula, shoulder acromioclavicular dislocation, shoulder dislocation.
* Cervical radiculopathy.
* Thoracic outlet syndrome.
* Restricted shoulder joint mobility due to stroke, spinal cord injury, or other factors.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain VAS | 90 days
  The intensity of the pain along a continuum from 'no pain' to 'worst pain' imaginable with visual analog scale.
ROM | 90 days
  Glenohumeral range of motion(ROM) of the affected shoulder.

SECONDARY OUTCOMES:
WHOQOL-BREF | 90 days
  A self-report questionnaire which assesses 4 domains of quality of life (QOL): physical health, psychological health, social relationships, and environment.
SPADI | 90 days
  Shoulder Pain and Disability Index (SPADI) is a 13-item patient completed instrument. Its categories include "pain" (5 items) and "disability" (8 items).
LDF | 90 days
  The Laser Doppler Flowmetry (LDF) is a widely used technology for monitoring microcirculatory status. Due to its excellent frequency response, ease of use, and tissue specificity, it is highly suitable for non-invasive microcirculatory examinations and be applied to detect microcirculation in frozen shoulder cases.
BPW | 90 days
  Blood pressure waveform(BPW) is a graphical representation or visual display of the changes in blood pressure over time measured through a radial artery pressure sensor.
PPG | 90 days
  Photoplethysmography(PPG), which is a non-invasive method used to detect blood volume changes in the microvascular bed of tissue

CONTACTS AND LOCATIONS:
Overall Officials: Ming Jen Wang, MD, Principal Investigator — Taipei City Hospital, Renai Branch, Chinese Medicine Department

IPD SHARING:
Plan to Share IPD: No